CLINICAL TRIAL: NCT04614714
Title: Nicotinamide Riboside and Milk Production in the NICU
Brief Title: Milk Volume Outcomes Following Oral Nicotinamide Riboside Supplementation in Mothers of Extremely Preterm Infants
Acronym: MOONRISE
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: ChromaDex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1557473
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Preterm Birth; Inadequate Milk Production
Keywords: Nicotinamide Riboside; milk volume; Neonatal intensive care unit; Galactagogue; Feasibility trial
MeSH Terms: conditions — Premature Birth | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide Riboside (NR) (Experimental): Mothers receive daily oral nicotinamide riboside chloride 250 mg supplementation per day for 14 days (+ 2 days extra capsule for loss or extending sample collection), from study Day 4 + 1 day [D4-5] to study Day 17 + 2 days [D17-19].
  Interventions: Other: Nicotinamide Riboside (NR)
- Placebo (Placebo Comparator): Mothers receive a daily oral placebo, microcrystalline cellulose 250 mg per day matched in appearance and schedule to the nicotinamide riboside supplement for 14 days (+ 2 days extra capsule for loss or extending sample collection), from study Day 4 + 1 day [D4-5] to study Day 17 + 2 days [D17-19].
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Nicotinamide Riboside (NR) — Mothers receive daily oral nicotinamide riboside chloride 250 mg supplementation per day for 14 days (+ 2 days extra capsule for loss or extending sample collection), from study Day 4 + 1 day [D4-5] to study Day 17 + 2 days [D17-19].
  Arms: Nicotinamide Riboside (NR)
Other: Placebo — Mothers receive a daily oral placebo, microcrystalline cellulose 250 mg per day matched in appearance and schedule to the nicotinamide riboside supplement for 14 days (+ 2 days extra capsule for loss or extending sample collection), from study Day 4 + 1 day [D4-5] to study Day 17 + 2 days [D17-19].
  Arms: Placebo

SUMMARY:
This study aims to evaluate the feasibility and effects of nicotinamide riboside (NR) supplementation in lactating mothers of infants expected to be hospitalized in the neonatal intensive care unit (NICU) for at least four weeks.

DETAILED DESCRIPTION:
An adequate supply of a mother's own milk plays a critical role in optimizing health outcomes for at-risk infants, such as preterm and medically or surgically complex term infants. Despite this, insufficient milk production disproportionately affects the mothers of these infants. In the United States, metoclopramide is the only drug approved by the FDA for off-label use as a galactagogue. Nicotinamide riboside (NR), a niacin precursor, has been shown in a murine model to support lean body composition in lactating dams while augmenting high-quality milk production and enhancing cognitive and physical development of pups. Human testing with NR has been limited to long-term safety and bioavailability measures. This study aims to assess the feasibility of NR supplementation in mothers whose infants are admitted to the NICU for at least 4 weeks.

To address this gap, this study will enroll a small cohort of mothers with infants, either born preterm (<32 weeks of gestation) or term infants with complex medical or surgical conditions, admitted to the NICU for at least four weeks.

This double-blinded, randomized, placebo-controlled pilot feasibility trial aims to investigate NR supplementation in mothers of infants who are hospitalized in the NICU for at least 4 weeks. The intervention period with maternal nicotinamide riboside supplementation/placebo and maternal milk, urine, and blood sampling will be 19 days, including an enrollment day.

We aim to establish the feasibility of conducting a supplementation study in mothers of hospitalized infants, with enrollment feasibility defined as enrolling ≥ 50% eligible mothers.

Secondary objectives include assessing feasibility metrics (supplement compliance, milk sample collection adherence, and withdrawal rates); protocol adherence; and the impact of nicotinamide riboside supplementation on milk volume, milk composition (including macro- and micronutrient composition, glycans, metabolites, lipidomics, and CCN3), and urinary metabolites. Remnant infant blood samples will be used to examine the relationship between infant feeding practices and neonatal insulin, glucose, and amino acid concentrations.

An optional component of the study is the collection of maternal blood to assess the impact of NR supplementation on the concentration of serum prolactin, AST, ALT, metabolites, and CCN3; plasma lipidomics; and whole blood concentration of NAD+ related precursors.

ELIGIBILITY:
Inclusion criteria are required to be met before or at enrollment:

Mothers who are 18 years or older.

Infants delivered at 24-32 weeks OR infants (any GA) that researchers anticipate will be hospitalized in the NICU for at least 4 weeks, including, but not limited to, infants with a diagnosis of gastroschisis, a cardiac defect, intestinal atresia, etc.

Infants born at the UC Davis Medical Center or transferred to the UC Davis Medical Center NICU within the first 7 days of life.

Mothers who attempted initial milk expression within 12 hours of delivery.

Mothers who attempted milk expression at least 6 times every 24 hours from 72 hours after delivery to the Enrollment Visit.

Mothers who have delivered at least 96 hours (4 days) prior to the Enrollment Visit.

Mothers who have experienced a level "3" on the OMPQ before starting the collection of their first 24-hour pooled milk sample (study days 0-3).

Mothers who plan to feed their infants breast milk for at least 3 months.

Mothers who were pregnant with one infant.

Mothers willing to refrain from tandem feeding (directly breastfeeding) another child during the study period.

Mothers willing to refrain from enrolling themselves in another intervention trial during the study period.

Mothers willing to express, weigh, record, and collect 24-hour pooled milk

Mothers willing to remove nipple piercings during the study period.

Mothers willing to refrain from using pseudoephedrine (often found in Sudafed, Theraflu, Claritin-D, etc.) during the study period.

Mothers willing to express milk 6 times or more every 24 hours, including at least once during the night, and with no more than 5 hours between milk expression sessions, during the study period.

Mothers willing to refrain from consuming non-study supplements that contain nicotinamide-riboside (or similar derivatives, including NMN) during the study period.

Mothers willing to refrain from consuming galactagogues during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 40 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrollment in a double-blind placebo-controlled supplementation trial in mothers of infants who are hospitalized. | Within 4 days post-delivery of the infant.
  Proportion of eligible mothers who consent to enrollment in the study.

SECONDARY OUTCOMES:
Difference in mean milk volume of expressed milk (mL) between NR and placebo | Volumes will be measured on study Day 0 + 3 days [baseline, pre-intervention], Study Day 10 ± 1 days [mid-intervention], and study Day 17 + 2 days [end of intervention].
  Comparison of total 24-hour expressed breast milk volume (in milliliters) between mothers receiving nicotinamide riboside and those receiving placebo.
Difference in human milk micronutrient concentrations between NR and placebo over time. | Milk samples will be collected on study Day 0 + 3 days [baseline, pre-intervention], Study Day 10 ± 1 days [mid-intervention], and study Day 17 + 2 days [end of intervention].
  Comparison of human milk micronutrient concentrations (Micrograms per liter (µg/L) or milligrams per liter (mg/L), depending on the element) between mothers receiving nicotinamide riboside and those receiving a placebo. Milk samples collected on study days will be analyzed using inductively coupled plasma mass spectrometry (ICP-MS) in a certified analytical laboratory.
Difference in amount and diversity of metabolites, including NAD+-related precursors and intermediates in milk between NR and placebo over time. | Milk samples will be collected on study Day 0 + 3 days [baseline, pre-intervention], Study Day 10 ± 1 days [mid-intervention], and study Day 17 + 2 days [end of intervention].
  NMR metabolomics will be used to compare the amount and diversity of metabolites, including NAD⁺-related precursors and intermediates (e.g., nicotinamide riboside, nicotinamide mononucleotide, nicotinamide, NAD⁺) between the NR group and the placebo from the milk samples collected on various study days.
Difference in human milk glycans (HMOs, glycoproteins, glycolipids) between NR and placebo over time. | Milk samples will be collected on study Day 0 + 3 days [baseline, pre-intervention], Study Day 10 ± 1 days [mid-intervention], and study Day 17 + 2 days [end of intervention].
  Comparison of human milk oligosaccharides (HMOs), glycoproteins, and glycolipids in milk samples collected on study days between NR and placebo groups using Nuclear magnetic resonance (NMR) spectroscopy-based metabolomics.
Difference in milk lipidomics in milk between NR and placebo over time. | Milk samples will be collected on study Day 0 + 3 days [baseline, pre-intervention], Study Day 10 ± 1 days [mid-intervention], and study Day 17 + 2 days [end of intervention].
  The difference in milk lipidomics between NR and placebo over time will be measured by Metabolon from samples collected on study days.
Difference in serum prolactin levels at day 18 and the change from the baseline between NR and placebo ( optional participation) | Study Day 3 + 1/-3 days [baseline] and Study Day 18 + 2/-1 days [end of study visit]
  Blood will be collected ( optional participation) on two occasions to look at the difference in serum prolactin levels between the Nicotinamide Riboside supplementation group and the placebo.
Difference in plasma lipidomics between NR and placebo(optional participation). | Study Day 3 + 1/-3 days [baseline] and Study Day 18 + 2/-1 days [end of study visit]
  Plasma samples will be analyzed using Metabolon's lipodomics platform to assess the effect of nicotinamide riboside ( NR) versus placebo on lipid metabolism. (Optional participation)
Difference in NAD+-related precursors and intermediates in K2 EDTA whole blood (optional participation) between NR and placebo over time. | Study Day 3 + 1/-3 days [baseline] and Study Day 18 + 2/-1 days [end of study visit]
  The difference in NAD+-related precursors and intermediates in K2 EDTA whole blood will be measured by NADMED between NR and placebo over time.
Difference in serum metabolites between NR and placebo (optional participation). | Study Day 3 + 1/-3 days [baseline] and Study Day 18 + 2/-1 days [end of study visit]
  Change in Serum NMR metabolites( analyzed by NMR-based metabolomics) will be compared between the nicotinamide riboside and placebo groups.
Feasibility metrics include supplement compliance, milk sample collection adherence, and withdrawal. | Total Day 18 + 2 days from the day of enrollment [Day 18-20]
  Proportion of enrolled mothers who adhere to the protocol without major deviations.
Difference in the concentration of CCN3 in milk between NR and placebo over time. | Milk samples will be collected on study Day 0 + 3 days [baseline, pre-intervention], Study Day 10 ± 1 days [mid-intervention], and study Day 17 + 2 days [end of intervention].
  Concentration of CCN3 in milk between NR and placebo over time using quantitative ELISA.
Difference in human milk protein, carbohydrate, and fat concentrations between NR and placebo over time. | Milk samples will be collected on study Day 0 + 3 days [baseline, pre-intervention], Study Day 10 ± 1 days [mid-intervention], and study Day 17 + 2 days [end of intervention].
  Differences in human milk protein, carbohydrate, and fat concentrations will be measured by Miris HMA™between NR and placebo over time.
Relationship between infant feeding practices and levels of plasma insulin, plasma amino acid, and plasma glucose in infant blood. | Day 1 of life- duration of NICU stay.
  Plasma insulin in an infant's blood will be measured from the remnant blood sample in the lab, if any, without having to do an extra blood draw from the infant for the study.
Relationship between infant feeding practices and levels of metabolites in infant blood. | Day 1 of life to the duration of NICU stay.
  The relationship between infant feeding practices will be compared with levels of metabolites measured by NMR metabolomics in infant blood from any remnant blood sample for the infant in the lab, without having to do an additional blood draw for the study.
Feasibility of supplement compliance and milk sample collection adherence, and withdrawal from the study | Study start to end of study
  Proportion of enrolled mothers who adhere to the protocol without major deviations.
Difference in maternal serum CCN3 between NR and placebo (Optional Participation) | Study Day 3 + 1/-3 days [baseline] and Study Day 18 + 2/-1 days [end of study visit]
  Difference in maternal serum CCN3 between NR and placebo at baseline and Day 18.

OTHER OUTCOMES:
Change in maternal weight (lbs.) | Study Day 3 ± 1 days [randomization, pre-intervention visit] and Study Day 18 + 2 days [end of study visit]
  This exploratory outcome measures change in maternal weight from baseline to the end of the study in participants receiving nicotinamide riboside versus placebo, measured using a calibrated digital scale at each study visit.
Outcome of growth parameters: Infant length (cm), weight(g), and head circumference ( cm). | Day 1 - Day 28
  This exploratory outcomes measure the changes in growth parameters (height, weight, and head circumference) using calculated z-scores (as measured by standard deviations from the mean, presented in percentages relative to the average for age).
NICU outcomes | Day 1 of life - end of NICU visit.
  NICU outcomes accessible in the EMR include morbidity, death, necrotizing enterocolitis, chronic lung disease, retinopathy of prematurity, and sepsis.
Difference in the concentration of urinary metabolites, including NAD+-specific metabolites as a proxy of NR supplementation, between NR and placebo over time. | Urine samples will be collected on two occasions, Study Day 3 ± 1 days [Randomization visit] and Study Day 18 + 2 days [End of study visit ]
  Urinary metabolites will be measured using nuclear magnetic resonance (NMR)-based metabolomics between the nicotinamide riboside (NR) and placebo groups.
Difference in serum biomarkers of liver function and calcium between NR and placebo (optional participation). | Study Day 3 + 1/-3 days [baseline] and Study Day 18 + 2/-1 days [end of study visit]
  Differences in serum biomarkers of liver function (AST/ALT) and calcium will be measured via a CMP between NR and placebo.
Diet, health, and anthropometric outcomes reported by mothers when their child turns 1, 2, and 3 years of age. | Day 1 of life to 3 years of age for the child.
  These will be obtained as a complete three-brief (10-15 minute) phone interviews when their child turns 1, 2, and 3 years old. Each call, conducted by study personnel after the child's annual well-child visit, will include a semi-structured survey about the child's diet, general health, and growth (weight, height, etc.). Participants will receive a $25 Amazon e-gift card for each completed interview (up to $75 total). Mothers may choose to complete one, two, or all three interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yang D, Wan Y. NR Supplementation During Lactation: Benefiting Mother and Child. Trends Endocrinol Metab. 2019 Apr;30(4):225-227. doi: 10.1016/j.tem.2019.02.004. Epub 2019 Feb 21. PMID 30797625
- [Result] Martens CR, Denman BA, Mazzo MR, Armstrong ML, Reisdorph N, McQueen MB, Chonchol M, Seals DR. Chronic nicotinamide riboside supplementation is well-tolerated and elevates NAD+ in healthy middle-aged and older adults. Nat Commun. 2018 Mar 29;9(1):1286. doi: 10.1038/s41467-018-03421-7. PMID 29599478
- [Result] Dollerup OL, Christensen B, Svart M, Schmidt MS, Sulek K, Ringgaard S, Stodkilde-Jorgensen H, Moller N, Brenner C, Treebak JT, Jessen N. A randomized placebo-controlled clinical trial of nicotinamide riboside in obese men: safety, insulin-sensitivity, and lipid-mobilizing effects. Am J Clin Nutr. 2018 Aug 1;108(2):343-353. doi: 10.1093/ajcn/nqy132. PMID 29992272
- [Result] Damgaard MV, Treebak JT. What is really known about the effects of nicotinamide riboside supplementation in humans. Sci Adv. 2023 Jul 21;9(29):eadi4862. doi: 10.1126/sciadv.adi4862. Epub 2023 Jul 21. PMID 37478182
- [Result] Trammell SA, Schmidt MS, Weidemann BJ, Redpath P, Jaksch F, Dellinger RW, Li Z, Abel ED, Migaud ME, Brenner C. Nicotinamide riboside is uniquely and orally bioavailable in mice and humans. Nat Commun. 2016 Oct 10;7:12948. doi: 10.1038/ncomms12948. PMID 27721479
- [Result] Conze D, Brenner C, Kruger CL. Safety and Metabolism of Long-term Administration of NIAGEN (Nicotinamide Riboside Chloride) in a Randomized, Double-Blind, Placebo-controlled Clinical Trial of Healthy Overweight Adults. Sci Rep. 2019 Jul 5;9(1):9772. doi: 10.1038/s41598-019-46120-z. PMID 31278280
- [Result] Ear PH, Chadda A, Gumusoglu SB, Schmidt MS, Vogeler S, Malicoat J, Kadel J, Moore MM, Migaud ME, Stevens HE, Brenner C. Maternal Nicotinamide Riboside Enhances Postpartum Weight Loss, Juvenile Offspring Development, and Neurogenesis of Adult Offspring. Cell Rep. 2019 Jan 22;26(4):969-983.e4. doi: 10.1016/j.celrep.2019.01.007. PMID 30673618
- [Result] Moller L, Crone KL, Mortensen N. [Brucellosis: 3 imported cases]. Ugeskr Laeger. 1985 Jul 1;147(27):2164-6. No abstract available. Danish. PMID 4060272
- [Result] Foong SC, Tan ML, Foong WC, Marasco LA, Ho JJ, Ong JH. Oral galactagogues (natural therapies or drugs) for increasing breast milk production in mothers of non-hospitalised term infants. Cochrane Database Syst Rev. 2020 May 18;5(5):CD011505. doi: 10.1002/14651858.CD011505.pub2. PMID 32421208
- [Result] Shen Q, Khan KS, Du MC, Du WW, Ouyang YQ. Efficacy and Safety of Domperidone and Metoclopramide in Breastfeeding: A Systematic Review and Meta-Analysis. Breastfeed Med. 2021 Jul;16(7):516-529. doi: 10.1089/bfm.2020.0360. Epub 2021 Mar 25. PMID 33769844
- [Result] Hussain NHN, Noor NM, Ismail SB, Zainuddin NA, Sulaiman Z. Metoclopramide for Milk Production in Lactating Women: A Systematic Review and Meta-Analysis. Korean J Fam Med. 2021 Nov;42(6):453-463. doi: 10.4082/kjfm.20.0238. Epub 2021 Nov 20. PMID 34871486
- [Result] Campbell-Yeo ML, Allen AC, Joseph KS, Ledwidge JM, Caddell K, Allen VM, Dooley KC. Effect of domperidone on the composition of preterm human breast milk. Pediatrics. 2010 Jan;125(1):e107-14. doi: 10.1542/peds.2008-3441. Epub 2009 Dec 14. PMID 20008425
- [Result] Grzeskowiak LE, Smithers LG, Amir LH, Grivell RM. Domperidone for increasing breast milk volume in mothers expressing breast milk for their preterm infants: a systematic review and meta-analysis. BJOG. 2018 Oct;125(11):1371-1378. doi: 10.1111/1471-0528.15177. Epub 2018 Mar 27. PMID 29469929
- [Result] Grzeskowiak LE, Wlodek ME, Geddes DT. What Evidence Do We Have for Pharmaceutical Galactagogues in the Treatment of Lactation Insufficiency?-A Narrative Review. Nutrients. 2019 Apr 28;11(5):974. doi: 10.3390/nu11050974. PMID 31035376
- [Result] Kwan SH, Abdul-Rahman PS. Clinical Study on Plant Galactagogue Worldwide in Promoting Women's Lactation: a Scoping Review. Plant Foods Hum Nutr. 2021 Sep;76(3):257-269. doi: 10.1007/s11130-021-00901-y. Epub 2021 Jul 22. PMID 34292494
- [Result] Zukova S, Krumina V, Buceniece J. Breastfeeding preterm born infant: Chance and challenge. Int J Pediatr Adolesc Med. 2021 Jun;8(2):94-97. doi: 10.1016/j.ijpam.2020.02.003. Epub 2020 Feb 6. PMID 34084879
- [Result] https://doi.org/10.1542/peds.2008-3441
- [Result] https://www.nadmed.com/wp-content/uploads/2025/03/RUO_Qualio-IFU-NAD-and-NADH-blood-v8.0-1.pdf
- [Result] Babey ME, Krause WC, Chen K, Herber CB, Torok Z, Nikkanen J, Rodriguez R, Zhang X, Castro-Navarro F, Wang Y, Wheeler EE, Villeda S, Leach JK, Lane NE, Scheller EL, Chan CKF, Ambrosi TH, Ingraham HA. A maternal brain hormone that builds bone. Nature. 2024 Aug;632(8024):357-365. doi: 10.1038/s41586-024-07634-3. Epub 2024 Jul 10. PMID 38987585